CLINICAL TRIAL: NCT07282652
Title: An Investigator-Initiated Study to Evaluate the Safety/Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of RAG-18 in Pediatric Patients With Duchenne Muscular Dystrophy
Brief Title: A Study to Evaluate the Safety and Tolerability of RAG-18 in Pediatric Patients With Duchenne Muscular Dystrophy
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Ractigen Therapeutics. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAG180101
Record Dates: First submitted 2025-11-17; First posted 2025-12-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RAG-18 (Experimental): The study will employ a dose-escalation design, enrolling participants into sequential cohorts for up to four planned dose levels. If the highest planned dose is well-tolerated, a decision to explore further dose escalation may be made based on the overall safety and risk-benefit evaluation.
  Interventions: Drug: RAG-18

INTERVENTIONS:
Drug: RAG-18 — RAG-18 is a therapeutic small activating RNA (saRNA) duplex molecule comprised of two partially chemically modified complementary oligonucleotide strands

SUMMARY:
This is an open-label, single-arm, dose-escalation trial to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy of RAG-18 in pediatric patients with Duchenne Muscular Dystrophy (DMD).

The study will enroll approximately 12 subjects into four cohorts to assess the safety and tolerability of ascending intravenous doses. Secondary objectives include characterizing the pharmacokinetics (PK)/pharmacodynamics (PD) profile and assessing exploratory efficacy through changes in muscle biomarkers, muscle composition, cardiac/pulmonary function, and motor performance. The decision to escalate to the next dose level will be based on a comprehensive safety evaluation of the preceding cohort.

ELIGIBILITY:
Inclusion Criteria:

1. In accordance with the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use - Good Clinical Practice (ICH-GCP) guidelines and local/national and/or Institutional Review Board (IRB)/Independent Ethics Committee (IEC) requirements, the participant and/or their legal guardian has signed the written informed consent form.
2. Aged 4-15 years old.
3. Male patient with Duchenne Muscular Dystrophy (DMD), able to provide a written diagnosis from a specialist and a verifiable genetic test report.
4. Able to undergo examinations required by the study protocol, such as muscle biopsy, Magnetic Resonance Imaging (MRI), and tests for motor and pulmonary function.
5. Any disease-related concomitant medications must be in compliance with the study's requirements.

Exclusion Criteria:

1. Prior treatment for Duchenne Muscular Dystrophy (DMD), regardless of whether the drug is marketed or not.
2. Body Mass Index (BMI) > 22 kg/m² or body weight ≥ 50 kg.
3. Unable to complete the motor function tests required by the protocol, including: North Star Ambulatory Assessment (NSAA), Time to Stand (TTSTAND), 4-Stair Climb (4SCV), and the 6-Minute Walk Test (6MWT).
4. Cardiac function at screening within the following ranges:

   * Left Ventricular Ejection Fraction (LVEF) < 55% as measured by Cardiac Magnetic Resonance (CMR).
   * QT interval corrected using Fridericia's formula (QTcF) > 450 ms at screening, or has additional risk factors for Torsades de Pointes.
5. Hematology and electrolyte parameters at screening within the following ranges:

   * Platelets < 100,000/μL.
   * Hemoglobin < 12 g/dL.
   * Absolute Neutrophil Count < 1500/μL.
   * Any serum calcium, potassium, sodium, magnesium, or phosphorus levels outside the clinically acceptable range for Duchenne Muscular Dystrophy (DMD) patients.
   * International Normalized Ratio (INR), Prothrombin Time (PT), Partial Thromboplastin Time (PTT), Activated Partial Thromboplastin Time (aPTT), or Fibrinogen outside the normal range.
6. History of medical conditions affecting liver function, with abnormal indicators within 28 days prior to the first dose.
7. Presence of severe cardiac, renal, or respiratory dysfunction, or other severe complications.
8. Allergy to the study drug or any of its components, or to Magnetic Resonance Imaging (MRI) contrast agents.
9. Receipt of a live (attenuated) vaccine within 28 days prior to the first dose of the study drug.
10. Use of any other investigational drug, whether for DMD or not, from 28 days prior to the first dose of the study drug until the end of the study.
11. Any reason that, in the investigator's opinion, would prevent the participant from fully participating in and completing the study, including inability to comply with study procedures or treatment, and other relevant medical or mental health conditions.
12. Presence of a severe concomitant condition or disease that, in the investigator's opinion, would place the participant at undue risk or interfere with the study, including but not limited to: known moderate or severe persistent asthma, a history of asthma in the past 2 years, or currently uncontrolled asthma of any classification (Note: participants with currently controlled intermittent asthma or controlled mild persistent asthma are permitted to enroll); requirement for oxygen therapy to maintain adequate blood oxygen saturation; history of Chronic Obstructive Pulmonary Disease (COPD) within 6 months prior to signing the Informed Consent Form (ICF).
13. Participant has an unstable systemic disease as judged by the investigator, including but not limited to severe hepatic, renal, respiratory, or metabolic diseases requiring medication.
14. Any other unspecified reason that, in the investigator's opinion, makes the participant unsuitable for enrollment.

Ages: 4 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Adverse Events (AEs) and Serious Adverse Events (SAEs) | From Baseline up to the end of the study (Day 169)
  To evaluate the safety profile of RAG-18 by recording the frequency, nature, and severity of all adverse events and serious adverse events observed during the study. The relationship of these events to the study drug will be assessed.

SECONDARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of RAG-18 | Day 1 and Day 85 (assessed at pre-dose, and multiple timepoints up to 168 hours post-dose)
  To evaluate the pharmacokinetic profile of RAG-18 after intravenous infusion.
Time to Maximum Observed Plasma Concentration (Tmax) of RAG-18 | Day 1 and Day 85 (PK samples collected at pre-dose and multiple timepoints up to 168 hours post-dose)
  To determine the time to reach the maximum observed plasma concentration of RAG-18.
Area Under the Plasma Concentration-Time Curve (AUC) of RAG-18 | Day 1 and Day 85 (PK samples collected at pre-dose and multiple timepoints up to 168 hours post-dose)
  To determine the total drug exposure over time by calculating the Area Under the Plasma Concentration-Time Curve (AUC).
Terminal Half-Life (t1/2) of RAG-18 | Day 1 and Day 85 (PK samples collected at pre-dose and multiple timepoints up to 168 hours post-dose)
  To determine the terminal elimination half-life of RAG-18 in plasma.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No